CLINICAL TRIAL: NCT02844504
Title: Neurophysiological Evaluation of Training Effect on Cancer-Related Weakness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Kessler Institute for Rehabilitation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-849-14; 5R01CA189665-02 (NIH)
Record Dates: First submitted 2016-06-23; First posted 2016-07-26 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer
Keywords: Fatigue; Breast cancer; Force; Motor imagery; Cancer Treatment
MeSH Terms: conditions — Breast Neoplasms; Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Intensity Exercise Training 1 (Experimental): Cancer survivors will receive low intensity handgrip exercise training.
  Interventions: Behavioral: Low Intensity Exercise Training 1
- Low Intensity Exercise Training 2 (Experimental): Cancer survivors will receive low intensity handgrip exercise training different than other arm.
  Interventions: Behavioral: Low Intensity Exercise Training 2
- Control (No Intervention): This group will receive no training.

INTERVENTIONS:
Behavioral: Low Intensity Exercise Training 1 — Subjects will perform handgrip exercise training at low intensity (20% maximal force) 5 times a week for 6 weeks (more details not provided to keep study blinded)
  Arms: Low Intensity Exercise Training 1
Behavioral: Low Intensity Exercise Training 2 — Subjects will perform a different handgrip exercise training at low intensity (20% maximal force) 5 times a week for 6 weeks (more details not provided to keep study blinded)
  Arms: Low Intensity Exercise Training 2

SUMMARY:
Breast cancer patients often suffer from long-term physical symptoms of weakness. In this study, investigators propose to compare how two different low intensity physical exercise training programs can improve handgrip strength for breast cancer patients with symptoms of weakness. Using brain imaging, the study will also investigate changes in brain structure, and muscle activity associated with handgrip.

DETAILED DESCRIPTION:
Participants will be randomized to either a no treatment group or one of two low intensity 6-week exercise training. Outcomes will be measured at baseline, post-intervention and 4 weeks post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 40-75 yrs
* Right handed, as determined by the Edinburgh Inventory (Oldfield, 1971)
* Proficient in English
* Must be available for the familiarization, and testing sessions

Exclusion Criteria:

* Symptoms for mild or severe depression as determined by a Patient Health Questionnaire (PHQ-8) score >14
* Significant cognitive impairments as defined by a score <28 in the Folstein Mini-Mental Screening Examination (MMSE, Folstein et al .1975).
* Participated in any type of motor imagery or strength training program in the last 5 years, or plan to start any motor imagery or physical strength training program for the 3 months duration of the study
* Neurological, psychiatric, musculoskeletal or other types of disorder that may affect participants sensorimotor function and cognitive abilities
* Current medication believed to affect cognitive/psychomotor function (i.e., opioid, analgesics, anxiolytics or antidepressants)
* History of alcohol, smoking, and drug abuse
* Any contraindication for MRI

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Hand grip force | Pretest (before training), Posttest (immediately after end of training), Retention test (4 weeks after end of training)
  Primary outcome will be used to compare pre to post change in maximum force contraction at the end of the 6-week intervention between groups.Similar comparison will be done between retention test (4 weeks after training) and posttest (immediately after training).

SECONDARY OUTCOMES:
Pre to Post changes of functional brain to muscle coupling at maximum handgrip contraction | Pretest (before training), Posttest (immediately after end of training), Retention test (4 weeks after end of training)
  Functional brain to muscle coupling will be measured by computing the EMG-EEG coherence before training, after training, and 4 weeks after end of intervention. Values will be compared between groups.
Pre to Post changes in EMG amplitude at maximum handgrip contraction | Pretest (before training), Posttest (immediately after end of training), Retention test (4 weeks after end of training)
  EMG of the right arm muscles will be assessed during maximum handgrip contraction before training, after training, and 4 weeks after end of intervention. Values will be compared between groups.
Pre to Post changes in Brain activity during maximum handgrip contraction | Pretest (before training), Posttest (immediately after end of training)
  functional magnetic resonance imaging will used to measure brain activity when subject performs maximum muscle handgrip contraction before training, after training. Values will be compared between groups.
Functional brain to muscle (EEG-EMG) phase coupling at low intensity handgrip muscle contraction. | Pretest (before training), Posttest (immediately after end of training), Retention test (4 weeks after end of training)
  Corticomuscular coherence between EEG signal from contralateral motor region and EMG signal from handgrip muscles will be computed while subjects perform handgrip contraction at 20% of their maximum force.Group x Time interaction will be measured.
EEG Brain connectivity during low intensity handgrip muscle contraction | Pretest (before training), Posttest (immediately after end of training)
  functional connectivity within the brain networks will be studied while subjects perform 20% of their maximum handgrip contraction. Group x Time interaction will be measured.
Fatigue sustained handgrip contraction task duration | Pretest (before training), Posttest (immediately after end of training), Retention test (4 weeks after end of training)
  Subjects will perform a sustained handgrip contraction task at 20% maximal force.The task duration (a measure of endurance) will be measured for each subject in the three groups, before and after training, and after 4 weeks of end of intervention. Group x Time interaction will be measured.
functional brain to muscle coupling during fatigue | Pretest (before training), Posttest (immediately after end of training), Retention test (4 weeks after end of training)
  EMG-EEG coherence will be studied when subjects get fatigue after performing a sustained muscle contraction task at 20% maximal force. Group x Time interaction will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Guang Yue, PhD, Principal Investigator — Kessler Foundation
Locations (2):
- United States (2):
  - Kessler Foundation, West Orange, New Jersey
  - Kessler Institute for Rehabilitation, West Orange, New Jersey

IPD SHARING:
Plan to Share IPD: No